CLINICAL TRIAL: NCT01752673
Title: The Visualization of Uncertainty in Clinical Diagnostic Reasoning for Pulmonary Embolism: a Randomized Controlled Trial.
Brief Title: The Visualization of Uncertainty in Clinical Diagnostic Reasoning for Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Ghazwan Altabbaa, Doctor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 23231
Record Dates: First submitted 2012-12-12; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Pulmonary Embolism; Diagnostic Uncertainty; Clinical Reasoning; Evidence Based Medicine; Visualization of Uncertainty
Keywords: randomized controlled study
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visualized pulmonary embolism computer task model (Experimental): This group of participants was presented and trained to use a visual representation of diagnostic pathway for pulmonary embolism. The design of this visual representation is based on Bayes theorem and cognition enhancing visual design principles.
  Interventions: Other: Visualized pulmonary embolism computer task model
- Didactic review pulmonary embolism lecture (Active Comparator): This group of participants was presented with a didactic lecture covering the diagnostic approach of pulmonary embolism.
  Interventions: Other: Didactic review lecture

INTERVENTIONS:
Other: Visualized pulmonary embolism computer task model — This group of participants was presented and trained to use a visual representation of diagnostic pathway for pulmonary embolism. The design of this visual representation is based on Bayes theorem and cognition enhancing visual design principles.
  Arms: Visualized pulmonary embolism computer task model
Other: Didactic review lecture — This group of participants was presented with a didactic lecture covering the diagnostic approach of pulmonary embolism.
  Arms: Didactic review pulmonary embolism lecture

SUMMARY:
Medical reasoning is a form of inquiry that examines the thought processes involved in making medical decisions. When physicians are faced with patients' symptoms or signs, their thought processes follow either direct shortcuts to suspect a diagnosis or go into a deeper and more analytic process to reach a diagnosis. The second pathway is less prone to biases and errors. This study explores whether the use of an interactive visual display of probabilities of pulmonary embolism generated from positive or negative test results will increase the adherence to evidence based guidelines in the diagnosis of pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Medical students, University of Calgary, in clerkship who finished at least 4 weeks of a block of medicine rotation at any hospital site.
* First year subspecialty or Internal Medicine residents.
* Practicing physicians in the subspecialties of Internal Medicine or Emergency Medicine.

Exclusion Criteria:

* Physicians in the subspecialty of Haematology or Respiratory

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Concordance with medical diagnostic reasoning pathway for pulmonary embolism. | Paper-based clinical case scenarios were completed within 2 hour after either intervention.
  Concordance with medical diagnostic reasoning pathway for a case presentation suggestive of pulmonary embolism will be reflected by whether participants are stopping prematurely or proceeding with diagnostic steps inappropriately.

SECONDARY OUTCOMES:
Time. | Paper-based clinical case scenarios were completed within 2 hour after either intervention.
  The overall time taken to solve each clinical scenario may give insight to which decision making process was predominant to solve each clinical scenario.

OTHER OUTCOMES:
Survey. | Survey was completed within 2 hours after completion of either intervention.
  The participants' responses to the satisfaction survey will provide feedback about the need for improvement or modification in interface of software

CONTACTS AND LOCATIONS:
Overall Officials: Ghazwan Altabbaa, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada